CLINICAL TRIAL: NCT00862316
Title: Outcome Analysis of the Oxford Unicompartmental Knee Arthroplasty With and Without the Assistance of a Computer Navigational Unit
Brief Title: Oxford Unicompartmental Knee Arthroplasty With and Without Navigational Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: Dartmouth General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA4
Record Dates: First submitted 2009-02-03; First posted 2009-03-16 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Knee Arthritis
Keywords: Eligible for Unicompartmental Knee Arthritis

ARMS (2):
- Computer Navigational Unit Assistance (Experimental): Oxford Unicompartmental Knee arthroplasty will be performed with the assistance of a computer navigational unit.
  Interventions: Device: Oxford Unicompartmental Knee
- Non- Computer Navigational Unit Assisted (Active Comparator): Oxford Unicompartmental Knee arthroplasty will be performed traditionally (without the assistance of a computer navigational unit).
  Interventions: Device: Oxford Unicompartmental Knee

INTERVENTIONS:
Device: Oxford Unicompartmental Knee — Knee Arthroplasty

SUMMARY:
The purpose of this study is to determine whether a computer navigational unit can improve operating time and consistency during Knee arthroplasty when compared to knee arthroplasty without a computer navigational unit.

DETAILED DESCRIPTION:
The ability to use a computerized navigational unit during knee arthroplasty can be a major benefit to surgeons that perform a small amount of knee arthroplasties. Navigational assistance can decrease surgery and anesthesia time as well as decreasing variation in posterior tibial slope and improved range of motion.

ELIGIBILITY:
Inclusion Criteria for the Oxford Knee

* symptomatic unicompartmental knee arthritis major surgery
* failed non operative treatment modalities
* willing and able to give informed consent
* skeletal maturity

Exclusion criteria for the Oxford Knee

* medical conditions that preclude general or spinal anesthetic
* ipsilateral knee avascular necrosis
* severe osteoporosis or osteopenia
* neuromuscular impairment
* ipsilateral knee infection

Patient day surgery criteria

* medically stable: an ASA category of 1 or 2
* close proximity to the hospital surgery performed for at least 36 hours
* good support system in place- someone able to stay with the patient for at least 36 hours immediately post-op.
* hemovac to be removed prior to discharge
* access to VON or other home care hospital approved services
* pain buster for pain control for 24 to 36 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Operative record | Immediately Post-Op
Visual Analogue for pain, activity, and patient satisfaction (VAS) | 1 year
American Knee Society Score (AKSS) | 1 year

SECONDARY OUTCOMES:
Oxford Knee 12 | 1 year
Western Ontario MacMaster(WOMAC) | 1 year
SF 12 | 1 year
Gait Belt Analysis | 1 year
Radiographic Output | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Venugopal, Dr., Principal Investigator — Dartmouth General Hospital
Locations (1):
- Dartmouth General Hospital, Dartmouth, Nova Scotia, Canada

REFERENCES:
- [Background] Svard UC, Price AJ. Oxford medial unicompartmental knee arthroplasty. A survival analysis of an independent series. J Bone Joint Surg Br. 2001 Mar;83(2):191-4. doi: 10.1302/0301-620x.83b2.10966. PMID 11284563
- [Background] Murray DW, Goodfellow JW, O'Connor JJ. The Oxford medial unicompartmental arthroplasty: a ten-year survival study. J Bone Joint Surg Br. 1998 Nov;80(6):983-9. doi: 10.1302/0301-620x.80b6.8177. PMID 9853489
- [Background] Price AJ, Webb J, Topf H, Dodd CA, Goodfellow JW, Murray DW; Oxford Hip and Knee Group. Rapid recovery after oxford unicompartmental arthroplasty through a short incision. J Arthroplasty. 2001 Dec;16(8):970-6. doi: 10.1054/arth.2001.25552. PMID 11740750
- [Background] Kreibich DN, Vaz M, Bourne RB, Rorabeck CH, Kim P, Hardie R, Kramer J, Kirkley A. What is the best way of assessing outcome after total knee replacement? Clin Orthop Relat Res. 1996 Oct;(331):221-5. doi: 10.1097/00003086-199610000-00031. PMID 8895642